CLINICAL TRIAL: NCT05859074
Title: A First-In-Human Phase I, Open Label, Safety and Tolerability Study of Escalating Multiple Doses of Intratumoral MQ710, a Multi-Transgene Expressing Modified Vaccinia Virus Ankara-Based Virotherapy, Alone and in Combination With the Systemic Checkpoint Inhibitor Pembrolizumab in Solid Tumors
Brief Title: A Study of MQ710 With and Without Pembrolizumab in People With Solid Tumor Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-278
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Squamous Cell Carcinoma; SCC - Squamous Cell Carcinoma; Basal Cell Carcinoma; BCC; BCC - Basal Cell Carcinoma; Melanoma; Merkel Cell Carcinoma; Sebaceous Carcinoma; Extramammary Paget Disease; Kaposi Sarcoma; Head and Neck Squamous Cell Carcinoma; HNSCC; Adnexal Carcinoma; Angiosarcoma; Cutaneous Neoplasm; Advanced Cancer; Metastatic Cancer; Refractory Cancer; Solid Tumor
Keywords: Cutaneous Squamous Cell Carcinoma; SCC - Squamous Cell Carcinoma; Basal Cell Carcinoma; BCC; Melanoma; Merkel Cell Carcinoma; Sebaceous Carcinoma; Extramammary Paget Disease; Kaposi Sarcoma; Head and Neck Squamous Cell Carcinoma; HNSCC; Adnexal Carcinoma; Angiosarcoma; Cutaneous Neoplasm; Advanced Cancer; Metastatic Cancer; Refractory Cancer; MQ710; Memorial Sloan Kettering Cancer Center; 22-278; Solid Tumor
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Basal Cell; Melanoma; Carcinoma, Merkel Cell; Adenocarcinoma, Sebaceous; Paget Disease, Extramammary; Sarcoma, Kaposi; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Skin Appendage; Hemangiosarcoma; Skin Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Group (Experimental): MQ710
  The dose levels will be escalated following a standard 3+3 dose escalation scheme.
  Interventions: Biological: MQ719
- Dose Expansion Group (Experimental): MQ710 + pembrolizumab
  Approximately 8 patients will be recruited into the dose expansion group for monotherapy dosing of MQ710. Approximately 12 patients will be recruited for dosing at the MTD/maximally administered dose established in combination with pembrolizumab.
  Interventions: Biological: MQ719; Drug: Pembrolizumab

INTERVENTIONS:
Biological: MQ719 — Patients will receive either multidose monotherapy with MQ710 or multidose combination therapy with MQ710 and pembrolizumab. The applicable dose of MQ710 will be injected directly into the patient's tumor (intratumorally), and standard dosing of pembrolizumab (200 mg) will be administered intravenously at a 3-week interval.
Drug: Pembrolizumab — Patients will receive either multidose monotherapy with MQ710 or multidose combination therapy with MQ710 and pembrolizumab. The applicable dose of MQ710 will be injected directly into the patient's tumor (intratumorally), and standard dosing of pembrolizumab (200 mg) will be administered intravenously at a 3-week interval.
  Arms: Dose Expansion Group

SUMMARY:
Participants of this study will have a diagnosis of a solid tumor cancer that has come back to its original location or spread beyond its original location (advanced), came back (relapsed) or worsened (refractory) after standard treatments, or no standard treatments are available for the participants' cancer. The purpose of this study if to find the highest dose of MQ710 that causes few or mild side effects in participants with a solid tumor cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Histologically or cytologically documented advanced or metastatic cancer that has relapsed from or is refractory to standard treatment in two lines of prior therapy in the advanced setting unless there are fewer than two FDA approved lines of therapy for the particular disease, or for which no standard treatment is available
* At least 2 tumors suitable for direct or ultrasound-guided injection defined as at least one cutaneous, subcutaneous, or nodal lesion or aggregate of lesions, ≥0.5 cm for any single lesion and cumulative lesion dimensions. One lesion must meet criteria for RECIST measurable disease if in Part 2. Note: One lesion will be biopsied (if possible)
* Mandatory initial screening biopsy

  a. For patients undergoing surgical excision/resection: i. Tumor deemed accessible and safe for biopsy by the Investigator ii. Willing to consent to biopsy and surgical procedure iii. Patient able to undergo surgical procedure and appropriate anesthesia b. For patients not undergoing surgical excision/resection to obtain mandatory screening biopsy: i. Tumor deemed accessible and safe for biopsy by the Investigator ii. Willing to consent to initial tumor biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients with no curative treatment options available including surgery and/or definitive radiation or patients in which these modalities are associated with significant morbidity
* Patients with advanced disease who have received and progressed on standard therapy or have disease for which there is no standard therapy or have contraindications to standard therapy

Part 1a: Patients with cutaneous squamous cell carcinoma (cSCC), basal cell carcinoma (BCC), melanoma, Merkel cell carcinoma, sebaceous carcinoma, extramammary Paget's disease, Kaposi sarcoma, HNSCC, adnexal carcinoma, and angiosarcoma, as well as patients with cutaneous neoplasms that are separate primaries with morbidity from multiple surgeries that have failed standard therapy. Any malignancy with superficial cutaneous or subcutaneous lesions or palpable lymph nodes may be eligible based on the discretion of the investigator.

* Part 2a: Patients with cutaneous squamous cell carcinoma (cSCC), basal cell carcinoma (BCC), melanoma, Merkel cell carcinoma, sebaceous carcinoma, extramammary Paget's disease, Kaposi sarcoma, HNSCC, adnexal carcinoma, and angiosarcoma, as well as patients with cutaneous neoplasms that are separate primaries with morbidity from multiple surgeries that have failed standard therapy. BCC will also be included, given that pembrolizumab has not been approved for this condition, although cemiplimab is approved.
* Parts 1b and 2b: Patients must have cSCC, Merkel cell carcinoma, melanoma, or head and neck squamous cell carcinoma. These patients should be refractory to anti-PD-1 therapy, with the exception of patients with HNSCC with PD-L1 expression <1.
* Parts 1a, 2a and 2b: Patients with BRAF-mutated melanoma should have received BRAF-targeted therapy.
* Predicted life expectancy of 3 months or more (in both Part 1 and Part 2)
* Participant or their legally authorized representative (LAR able to provide written informed consent to participate
* Ability to comply with study procedures in the Investigator's opinion
* Adequate renal function as defined by Cr <2 mg/dL
* Adequate hepatic function

  1. Serum bilirubin ≤1.5 x ULN
  2. AST and ALT ≤2.5 ULN (no liver mets)
  3. AST and ALT ≤5.0 ULN (for patients with liver mets)
* Adequate bone marrow and hematologic function

  1. Coagulation function adequate (PT and aPTT within x1.5 ULN)
  2. Platelets ≥ 75,000/mm^2
  3. ANC ≥ 1000/uL
* Females of child-bearing potential must have a negative pregnancy test within 14 days prior to enrollment and on day of treatment. All patients must agree to use adequate contraception prior to study entry, for the duration of study participation, and up to 90 days after the last dose of MQ710
* Part 2 only: at least one measurable site of disease according to RECIST criteria
* Prior non-immunotherapy, anti-tumor treatment including endocrine, chemical/radiotherapy, targeted therapy, or major surgery (but not anti-PD1/- L1 therapies) was discontinued for more than 4 weeks prior to enrollment
* Patients who have failed prior anti-PD1/-PDL1 may be included. Washout of anti-PD1/-PDL1 at least 3 weeks prior to initiation of therapy in Part 1a and 2a. No washout period is required for Part 1b and 2b.

Exclusion Criteria:

* Splenectomy
* Active infections requiring antibiotics, physician monitoring or recurrent fevers (>38.0 ℃) associated with a clinical diagnosis of active infection
* Acute or chronic active viral disease or positive test for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV) with CD4 count <100mg/m3, or received treatment with antivirals or nucleoside analogs such as those used in the treatment of hepatitis B (e.g. lamivudine, adefovir, tenofovir, telbivudine, entecavir), ribavirin, cidofovir, diaminopurine analogs, methyladenosine analogs, or interferon alpha within 4 weeks of initiation of study treatment .a. Patients with HIV are allowed on study if CD4 count is >100 cells/mm3.
* Incomplete recovery from surgery, incomplete healing of an incision site
* Any of the following in the 3 months before the first dose of study treatment: Grade 3 or 4 gastrointestinal bleeding/haemorrhage (unless due to resected tumour), treatment-resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thrombo-embolic event, history or evidence of haemoptysis or menorrhagia
* History of myocardial infarction, myocarditis, congestive heart failure (as defined by New York Heart Association Functional Classsification III or IV), unstable angina, serious uncontrolled cardiac arrhythmia,or significant cardiovascular or cerebrovascular event in the 6 months before the first dose of study treatment
* Uncontrolled infection within 6 months prior to study entry.
* History of significant bleeding requiring hospitalization in the 12 months before the first dose of study treatment
* Treatment with PD-1/programmed death ligand (PD-L1), cytotoxic T-lymphocyte associated protein 4 (CTLA-4), or any other (including experimental) immune checkpoint inhibitor or immune-stimulatory treatment in the 3 weeks before the first dose of study treatment
* Prior chemotherapy, radiotherapy, biological cancer therapy (not including anti-PD1/-L1 immunotherapies), targeted therapy, investigational drug, or major surgery 28 days prior to enrollment or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment with the exception of grade 2 or better for alopecia and neuropathy.
* Has known active CNS metastases and/or carcinomatous meningitis
* Received live vaccine within 28 days prior to enrollment
* Patient is pregnant or breast-feeding, or expecting to conceive or father children within the duration of the trial
* Patients with tumor that directly contacts, encases or penetrates a major blood vessel, pericardium, gastrointestinal tract, or other hollow organs that may lead to perforation due to tumor necrosis
* Patients at risk of airway compromise in the event of post-injection tumor swelling/inflammation based on investigator judgement
* History or evidence of autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)
* History of chronic liver disease or evidence of hepatic cirrhosis
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia, active interstitial lung disease (ILD) requiring treatment with systemic steroids
* Baseline pulse oximetry less than 92% on room air
* History of re-irradiation to a field which includes the carotid arteries
* History of leukemia: ALL and CLL (patients with a history of aggressive lymphomas in remission or patients with a history of allogeneic stem cell transplants are eligible if no longer on immunosuppressive therapy and without evidence of GvHD)
* Current use of steroids such as prednisone 10 mg/daily or greater (or its equivalent) or immunosupressants within 2 weeks of initiation of study treatment
* Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results
* Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
* Known allergy to MQ710 transgene products or formulation.
* Patient requires anticoagulation therapy, such as warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2028-05-04 (Estimated); Study Completion 2028-05-04 (Estimated)

PRIMARY OUTCOMES:
Safety of MQ710 by review of AEs and SAEs | Up to 2 years
  Review the safety and tolerability of MQ710 by review of AE's and SAE's by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lara Dunn, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org